CLINICAL TRIAL: NCT04369040
Title: Comparison of Two Ventilation Systems in Laryngeal Surgery: High-flow Nasal Oxygen Therapy and Laryngeal Micro-catheter With the Ventinova Technique
Brief Title: Comparison of Two Ventilation Methods for Micro-Laryngeal Surgery
Acronym: Ventinova ORL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty of recruiting and changing anesthesia methods
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_0016
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Laryngeal Disease
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-flow nasal oxygen therapy (Other): Ventilation with High-flow nasal oxygen therapy
  Interventions: Device: High-flow nasal oxygen therapy using a specific nasal cannula
- Flow Controlled Ventilation (Experimental): Ventilation with laryngeal tri-tube with Flow Controlled Ventilation technique
  Interventions: Device: Flow Controlled Ventilation using a laryngeal tri-tube

INTERVENTIONS:
Device: High-flow nasal oxygen therapy using a specific nasal cannula — Patient in this arm will received high-flow nasal oxygen therapy ventilation during the ENT surgery
  Arms: High-flow nasal oxygen therapy
Device: Flow Controlled Ventilation using a laryngeal tri-tube — Patient in this arm will received a laryngeal tri-tube ventilation during the ENT surgery
  Arms: Flow Controlled Ventilation

SUMMARY:
Single-center, randomized study, comparing two methods of oxygenation on 80 patients

DETAILED DESCRIPTION:
This study is a single-center, randomized study, comparing two methods of oxygenation during micro-laryngeal surgery performed under general anesthesia and myorelaxation: high-flow nasal oxygen therapy (HFNO) or Flow Controlled Ventilation (FCV) using a laryngeal tri-tube. The study population will be composed of 80 patients, aged over 18 and under 80.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18 and under the age of 80
* Patient to benefit from micro-laryngeal ENT surgery under general anesthesia and myorelaxation with an estimated duration which does not exceed 30 minutes
* Having signed a consent form
* Being affiliated with a Health Insurance plan.

Exclusion Criteria:

* Pregnant or lactating patient
* Patient with a weight <40 kg
* Obese patient (BMI> 30)
* Patient with foreseeable intubation difficulty
* Patient maintained under general anesthesia postoperatively
* Surgery requiring time by surgical laser
* Surgery involving the use of an active electrosurgical electrode in the immediate area of the electrosurgical device or electrode
* Predictable surgery longer than 30 minutes
* Being deprived of liberty or under guardianship.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Compare the percentage of patients having oxygen desaturation during the procedure or a PaCO2 > 65 mmHg at its end with both methods (high-flow nasal oxygen therapy and the use of FCV modality via a laryngeal tri-tube). | 1 day (during surgery)
  % of patients having an oxygen desaturation (SpO2<92%) during the procedure OR a PaCO2 > 65 mmHg at its end

SECONDARY OUTCOMES:
Evaluate the duration of oxygen therapy before desaturation in the two groups | 1 day (during surgery)
  Delay before oxygen desaturation (SpO2<92%) during the procedure
Evaluate the quality of the visualization of the laryngeal region in the two groups | 1 day (during surgery)
  Percentage of glottic opening (POGO) score at laryngoscopy
Evaluate the time-PaCO2 (partial pressure of carbon dioxide) relationship according to the techniques | 1 day (during surgery)
  PaCO2 (partial pressure of carbon dioxide) at the end of the procedure
Evaluate the possibility of a decrease in FiO2 (Fraction of inspired oxygen) | 1 day (during surgery)
  Minimal inspired fraction of oxygen during the procedure
Evaluate the incidence of atelectasis | 1 day (during surgery)
  Incidence of atelectasis on a postoperative chest X ray
Evaluate the time taken to resume spontaneous ventilation and wake up when the anesthetic agents are stopped | 1 day (during surgery)
  Delay between the end of administration of anesthetic drugs and return to spontaneous ventilation
Evaluate the incidence of postoperative complications on day 1 in relation to the technique | 1 day
  Incidence of postoperative complications at day 1 after the surgery
Evaluate the incidence of postoperative complications on day 7 in relation to the technique | 7 days
  Incidence of postoperative complications up to day 7

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, Dr, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No